CLINICAL TRIAL: NCT01057823
Title: Environment and Perceived Control: Improving Sleep in Hospitalized Older Patients
Brief Title: Understanding Sleep in Hospitalized Older Patients
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 16685B; 1K23AG033763-01 (NIH)
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Sleep Deprivation; Sleep Fragmentation
Keywords: aged; sleep deprivation; actigraphy; ambulatory monitoring
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Inpatient Elders Age 50 and up: The study population is community-dwelling ambulatory patients age 50 or above hospitalized on the University of Chicago general medicine service. Exclusion criteria include: (1) transfer from the ICU or another hospital; (2) cognitively impaired; (3) not ambulatory; (4) residents of a nursing home or skilled nursing facility; (5) on bedrest; (6)documented sleep disorder in their medical history (i.e. obstructive sleep apnea, narcolepsy, etc).

SUMMARY:
The overall goal of this research is to elucidate how environmental, healthcare, and patient-level factors and patients' level of perceived control impact sleep duration and quality in hospitalized older patients and to assess whether better in-hospital sleep is associated with improved physical activity and health outcomes.

We hypothesize that environment, healthcare disruptions and patient symptoms will be significantly associated with objective and subjective sleep duration and sleep quality in hospitalized older patients.

We also hypothesize that a high level of perceived control will be associated with improved sleep duration and quality in hospitalized older patients.

We further hypothesize that shorter sleep duration and quality in hospitalized older adults will be associated with adverse health outcomes, namely higher blood pressure and blood sugar.

DETAILED DESCRIPTION:
This research can lead to a better understanding of the effects of inpatient sleep on health outcomes for hospitalized older patients and can help inform the design and evaluation of interventions designed to improve sleep in hospitalized older patients. This work can also form the foundation for understanding the longer term health effects of inpatient sleep loss for older patients that are potentially modifiable.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or above
* Hospitalized on General Medicine service
* Ambulatory
* Community Dwelling
* MMSE >17

Exclusion Criteria:

* transfer from the ICU or another hospital
* cognitively impaired
* not ambulatory
* residents of a nursing home or skilled nursing facility
* on bedrest
* documented sleep disorder in their medical history

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community-dwelling ambulatory patients age 50 or above hospitalized on the University of Chicago general medicine service.
Sampling Method: Probability Sample
Enrollment: 771 (Actual)
Dates: Start 2010-01; Primary Completion 2019-07-19 (Actual); Study Completion 2020-07-19 (Actual)

PRIMARY OUTCOMES:
Sleep will be measured using subjective reports (Karolinska Sleep Diary on Daily Sleep Assessment). | January 2010-January 2015

SECONDARY OUTCOMES:
Sleep will also be measured objectively using actigraphy. | January 2010-January 2015

CONTACTS AND LOCATIONS:
Overall Officials: Vineet M Arora, MD, MA, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Result] Arora VM, Chang KL, Fazal AZ, Staisiunas PG, Meltzer DO, Zee PC, Knutson KL, Van Cauter E. Objective sleep duration and quality in hospitalized older adults: associations with blood pressure and mood. J Am Geriatr Soc. 2011 Nov;59(11):2185-6. doi: 10.1111/j.1532-5415.2011.03644.x. No abstract available. PMID 22098044
- [Result] Yoder JC, Staisiunas PG, Meltzer DO, Knutson KL, Arora VM. Noise and sleep among adult medical inpatients: far from a quiet night. Arch Intern Med. 2012 Jan 9;172(1):68-70. doi: 10.1001/archinternmed.2011.603. No abstract available. PMID 22232151
- [Result] Adachi M, Staisiunas PG, Knutson KL, Beveridge C, Meltzer DO, Arora VM. Perceived control and sleep in hospitalized older adults: a sound hypothesis? J Hosp Med. 2013 Apr;8(4):184-90. doi: 10.1002/jhm.2027. Epub 2013 Mar 18. PMID 23504939
- [Derived] DePietro RH, Knutson KL, Spampinato L, Anderson SL, Meltzer DO, Van Cauter E, Arora VM. Association Between Inpatient Sleep Loss and Hyperglycemia of Hospitalization. Diabetes Care. 2017 Feb;40(2):188-193. doi: 10.2337/dc16-1683. Epub 2016 Nov 30. PMID 27903614